CLINICAL TRIAL: NCT00307892
Title: A Randomised, Double- Blind, Placebo Controlled, Clinical Trial to Assess the Efficacy of the Homeopathic Medication TRAUMEEL S in Reducing Pain After Arthroscopy
Brief Title: Traumeel S for Reduction of Post Operative Pain Following Arthroscopy
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Inability to recruit patients
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Menachem Oberbaum, MD, Shaare Zedek Medical Center, Jerusalem, Israel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Arth 06 CTIL
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-10

CONDITIONS: Post-operative Pain
Keywords: Homeopathy; Traumeel S; Arthroscopy; Pain management; Post-operative pain following arthroscopy
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Eating

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Active Comparator): TRAUMEEL S
  Interventions: Drug: Traumeel S: intra-operative irrigation + oral ingestion
- B (Placebo Comparator): comparable placebo remedy (injection and oral)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Traumeel S: intra-operative irrigation + oral ingestion — homeopathic remedy
  Arms: A
Drug: Placebo — placebo remedy
  Arms: B

SUMMARY:
The perception of pain is a complex process that is not yet fully understood. With outpatient knee arthroscopy becoming standard of care, postoperative pain management has become increasingly important in caring for patients. Traumeel S is a homeopathic complex widely used in German-speaking Europe for orthopedic pain and inflammation. It contains a mixture of medicinal plants and minerals, all highly diluted. In some recent studies, Traumeel has shown anti-inflammatory and analgesic activity.

In this study, the efficacy of Traumeel S will be compared with placebo in reducing pain during the first 48 hours after arthroscopy. Also compared will be 6 day pain levels, analgesic consumption, quality of life, post operative knee function, quadriceps atrophy and safety.

The study design is double blind RCT. 98 patients, aged 18-40 and undergoing arthroscopic meniscectomy or chondroplasty will be enrolled in the trial. Patients will be randomized to receive either intraoperative join irrigation with Traumeel S and oral treatment with Traumeel S, or placebo irrigation and oral ingestion. Patients will continue to take active or placebo medication for 6 days. Pain will be recorded daily by the patient in the patient diary using an 11-point numerical rating score (NRS-11. Patients will also record daily consumption of primary and "rescue" analgesics. Range of motion (RoM) will be measured on days 6 and 30 post-operatively, and the Lysholm knee scale and circumference of thigh above patella will be measured at 30 days. All these measures will be compared with baseline. Patients will be contacted daily by the research assistant to encourage compliance and to record their daily NRS and analgesic consumption in the CRF.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex undergoing unilateral arthroscopy for menisectomy or chondroplasty, w/o ligament reconstruction .
* Age 18 - 40 years.
* Meeting none of exclusion criteria.

Exclusion Criteria:

* Participation in another clinical trial within 4 weeks prior to enrollment.
* Inability to comply with the study protocol.
* Impossibility to be reached during the whole follow-up period (7 days post operative)
* Refused to give oral consent to the telephone interviews
* Previous arthroscopy on ipsilateral knee.
* Current use of analgesia for any other reason except for the knee complaint.
* Any disease considered to inhibit wound healing (e.g. Diabetes mellitus, Berger, any PVD, DVT).
* Known sensitivity to dipyrone or diclofenac

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Degree of pain at rest, as recorded daily by the patient and by the study assistant in the CRF, using a 11 point (0-10) numerical rating score (NRS-11), during the first two post operative days. | 30d

SECONDARY OUTCOMES:
Degree of pain at rest, as recorded daily by the patient and by the study assistant in the CRF, using a 11 point (0-10) numerical rating score (NRS-11), during the six post operative days. | 30d
Total amount of primary oral analgesic tablets ingested, as reported by the patient and the study assistant in the CRF from Day 0 to Day 5 (six days), using a discrete scale. | 30d
Number of days on which oral rescue analgesic treatment was required, if any, as reported by the patient and the study assistant in the CRF, from Day 0 to Day 5 (six days) using a discrete scale. | 6d
Degree of pain upon performance of RoM on days 5 and 30 postoperatively as compared with baseline, using a 11 point (0-10) numerical rating score (NRS), along a discrete scale. | 30d
Knee function as measured by difference in RoM at 5 and 30 days postoperatively, as compared with baseline, on a continuous scale. | 30d
Degree of atrophy of quadriceps, as measured by difference in circumference of thigh 15 cm proximal to the upper pole of the patella with knee in full extension on 30 days post-operatively, as compared with baseline, on a continuous scale. | 30d
Difference in disease-related QoL, as measured by the difference in Lysholm knee score on 30 days post operatively as compared with baseline . | 30d
Occurrence of adverse events. | 30d

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Oberbaum, M.D., Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Dept. of Orthopedic Surgery, Shaare Zedek Medical Center, Jerusalem, Israel